CLINICAL TRIAL: NCT03724747
Title: A Phase 1, Open-label, First-in-human, Multi-center, Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of a Thorium-227 Labeled Antibody-chelator Conjugate, BAY 2315497 Injection Alone, and in Combination With Darolutamide (BAY 1841788), in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Study to Evaluate the Safety, Tolerability,Pharmacokinetics, and Antitumor Activity of a Thorium-227 Labeled Antibody-chelator Conjugate Alone and in Combination With Darolutamide, in Patients With Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19445; 2018-001490-25 (EudraCT Number)
Record Dates: First submitted 2018-10-23; First posted 2018-10-30 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Castration Resistant Prostate Cancer (mCRPC)
Keywords: Metastatic castration resistant prostate cancer, thorium-227, targeted alpha therapy,PSMA
MeSH Terms: interventions — BAY 2315497

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- BAY2315497 dose escalation (Experimental): The thorium-227 dose will be escalated in a step-wise fashion to the MTD, according to a predefined dose escalation scheme. The total antibody dose of 50 mg will be evaluated first; on the basis of emerging clinical data, doses within the range of 20-100 mg may be investigated.
  Interventions: Drug: BAY2315497 Injection
- BAY2315497 dose escalation in combination with darolutamide (Experimental): The thorium-227 dose will be escalated in a step-wise fashion to the MTD, according to a predefined dose escalation scheme. In addition, Darolutamide oral dosing at the approved dose of twice daily 600 mg will be initiated 14 days prior to the first BAY2315497 Injection dose on Day 1 of the first cycle. Daily darolutamide dosing will continue throughout the entire BAY2315497 Injection treatment period until withdrawal criteria from study treatment period are met.
  Interventions: Drug: BAY2315497 Injection; Drug: Darolutamide(BAY1841788)
- BAY2315497 dose expansion:Dose regimen 1 (Experimental): The thorium-227 and total antibody doses, as well as the treatment regimen, will be selected for expansion on the basis of the safety, PK and overall benefit risk profile of BAY2315497 Injection, observed in the course of the dose escalation.
  Interventions: Drug: BAY2315497 Injection
- BAY2315497 dose expansion:Dose regimen 2 (Experimental): The thorium-227 and total antibody doses, as well as the treatment regimen, will be selected for expansion on the basis of the safety, PK and overall benefit risk profile of BAY2315497 Injection, observed in the course of the dose escalation.
  Interventions: Drug: BAY2315497 Injection

INTERVENTIONS:
Drug: BAY2315497 Injection — BAY 2315497 Injection comprises 3 components: the PSMA-specific monoclonal antibody (mAb), the mAb-chelator conjugate, and the thorium-227 labeled mAb-chelator conjugate. BAY 2315497 Injection will be administered on Day 1 of each treatment cycle.
Drug: Darolutamide(BAY1841788) — 600 mg (2 X 300 mg tablets), twice daily with food, equivalent to a total daily dose of 1200 mg.
  Arms: BAY2315497 dose escalation in combination with darolutamide

SUMMARY:
The study medication (BAY 2315497 Injection) is a thorium-227 labeled immuno-conjugate, specific for the prostate-specific membrane antigen (PSMA), which will be evaluated in patients with metastatic castration resistant prostate cancer. In this study, this investigational medication will be administered to patients for the first time. The primary objective of the study is to define the safety and tolerability profile and Maximal Tolerated Dose (MTD) of BAY2315497 Injection alone, or in combination with darolutamide. The secondary objectives are to determine the recommended dose for further clinical development of BAY2315497 Injection alone, or in combination with darolutamide and to investigate how the study drug is distributed and cleared from the body.

ELIGIBILITY:
Inclusion Criteria

* Ability to understand and sign an approved informed consent form.
* Male adult patients (≥ 18 years of age).
* ECOG PS of 0 or 1.
* Life expectancy ≥ 6 months.
* Histological, pathological and/or cytological confirmation of adenocarcinoma of the prostate without small cell or neuroendocrine features.
* Previous treatment with at least one novel androgen axis drug (NAAD) (e.g. enzalutamide and/or abiraterone).
* Patients must have prior orchiectomy and/or ongoing androgen deprivation therapy and a castrate level of serum testosterone (<50 ng/dL or <1.7 nmol/L).
* Previous treatment with at least 1, but no more than 2 previous - taxane regimens. A taxane regimen is defined as a minimum exposure of 2 cycles of a taxane. If a patient has received only 1 taxane regimen, he is eligible, if refuses to receive a second taxane regimen, or is considered unsuitable to receive a second taxane regimen (e.g. intolerance).
* Documented progression of mCRPC, as defined according to the Prostate Cancer Working Group 3 (PCWG3) guidelines.
* Adequate bone marrow, liver, and renal function, as assessed by the following laboratory requirements, to be conducted within 14 days before start of study drug administration:

  * Hemoglobin > 9.0 g/dL
  * Absolute neutrophil count (ANC) > 1500/mm3
  * White blood cell (WBC) count > 3000/mL
  * Platelet count > 100,000 /mm*3
  * Total bilirubin < 1,5 x upper limit of normal (ULN) (except if confirmed history of Gilbert's disease)
  * ALT and AST ≤ 2.5 x ULN
  * Serum creatinine ≤ 1.5 X ULN and glomerular filtration rate (GFR ≥ 45 mL/min/1.73 m2, according to the MDRD (Modified Diet in Renal Disease) abbreviated formula.
* Patients with partners of childbearing potential must be willing to use highly effective methods of birth control for the time period between the first administration of BAY 2315497 Injection to at least 6 months after the last administration of the study drug.
* In the darolutamide BAY2315497 Injection combination escalation arm, patients at sites performing the PSMA and FDG PET/CTs should be able to tolerate the 3 radiotracer injections and the 3 whole body PET/CT scans.

Exclusion Criteria

* Diffuse bone or bone-marrow involvement (i.e. "superscan").
* Spinal cord compression or known brain metastases.
* Known incompatibility to CT/MRI, bone scan or uncontrolled pain, which results in patient's lack of compliance with the CT/MRI and bone scan required for PCWG3 tumor assessment.
* Clinically significant heart disease, as evidenced by myocardial infarction, arterial thrombotic events in the past 6 months, severe or unstable angina, or uncontrolled cardiovascular history.
* Patients known to be affected by genetic defects linked to radiation Hypersensitivity.
* Known history of myelodysplastic syndrome (MDS) / leukemia or with features suggestive of MDS/AML at any time point.
* Concurrent or active cancer within the last 2 years with a distinct primary site or histology from the cancer being evaluated in this study, with the exception of cancer types with less than 30% likelihood of recurrence.
* Known allergies, hypersensitivity, or intolerance to the study drug including excipients, or to contrast agents used in the diagnostic or exploratory imaging procedures required per protocol.
* Any infection of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 Grade ≥ 2.
* Known human immunodeficiency virus (HIV) infection.
* Patients who have an active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection requiring treatment.
* Serious, non-healing wound, ulcer, or bone fracture.
* Any systemic anti-neoplastic therapy (e.g. chemotherapy, immunotherapy or biological therapy [including monoclonal antibodies], PARP inhibitors) within at least 30 days prior to day of randomization (except for Luteinizing Hormone-releasing Hormone [LHRH] or Gonadotropin-releasing Hormone [GnRH]).
* Previous high-dose chemotherapy, needing hemopoietic stem cell rescue, is prohibited.
* Prior major surgery (excluding prostatic biopsies) must be at least 12 weeks prior to study entry.
* Previous treatment with therapeutic PSMA-targeted agents.
* Previous treatment with radium-223 dichloride or other radiopharmaceuticals, including but not limited to strontium-89 or samarium-153.
* Prior definitive radiotherapy completed less than 6 weeks before start of the study drug administration
* Inability to swallow oral medications
* A gastrointestinal disorder or procedure which is expected to interfere significantly with absorption of darolutamide

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of BAY2315497 injection | Cycle 1 (42 days)
  The maximum dose at which the incidence of DLTs occurring during Cycle 1 is below 30%.
Maximum tolerated dose (MTD) of BAY2315497 injection in combination with darolutamide | Cycle 1 (42 days)
  The maximum dose at which the incidence of DLTs occurring during Cycle 1 is below 30%.

SECONDARY OUTCOMES:
Recommended dose for further clinical development of BAY2315497 injection | Up to 6 cycles (each cycle is 42 days, a maximum of 3 additional treatment cycles may be administered in case a favorable benefit risk profile is documented)
  The dose / regimen recommended for further clinical development will be defined after evaluation of the safety, PK and overall clinical data, collected in cycle 1 and subsequent cycles, in the dose escalation and dose expansion parts of the study.
Maximum observed concentration (Cmax) of thorium of BAY2315497 Injection | Cycle 1 (From day 1 to 43)
Area under the curve from time of dosing to 42 days after dosing [AUC(0-42)] days of thorium of BAY2315497 Injection | Cycle 1 (From day 1 to 43)
Cmax of radium of BAY2315497 Injection | Cycle 1 (From day 1 to 43)
AUC(0-42) days of radium of BAY2315497 Injection | Cycle 1 (From day 1 to 43)
Cmax of total antibody of BAY2315497 Injection | Cycle 1 (From day 1 to 43)
AUC(0-42) days of total antibody of BAY2315497 Injection | Cycle 1 (From day 1 to 43)
Recommended dose for further clinical development of BAY2315497 injection in combination with darolutamide | Up to 6 cycles (each cycle is 42 days, a maximum of 3 additional treatment cycles may be administered in case a favorable benefit risk profile is documented)
  The dose / regimen recommended for further clinical development will be defined after evaluation of the safety, PK and overall clinical data, collected in cycle 1 and subsequent cycles, in the dose escalation and dose expansion parts of the study.
Maximum observed concentration (Cmax) of thorium of BAY2315497 Injection in combination with darolutamide | Cycle 1 (From day 1 to 43)
Area under the curve from time of dosing to 42 days after dosing [AUC(0-42)] days of thorium of BAY2315497 Injection in combination with darolutamide | Cycle 1 (From day 1 to 43)
Cmax of radium of BAY2315497 Injection in combination with darolutamide | Cycle 1 (From day 1 to 43)
AUC(0-42) days of radium of BAY2315497 Injection in combination with darolutamide | Cycle 1 (From day 1 to 43)
Cmax of total antibody of BAY2315497 Injection in combination with darolutamide | Cycle 1 (From day 1 to 43)
AUC(0-42) days of total antibody of BAY2315497 Injection in combination with darolutamide | Cycle 1 (From day 1 to 43)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Tulane Medical Center, New Orleans, Louisiana
  - GU Research Network, LLC, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- HUS, Meilahden sairaala, Helsinki, Finland
- Royal Marsden NHS Trust (Surrey), Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Hammer S, Hagemann UB, Zitzmann-Kolbe S, Larsen A, Ellingsen C, Geraudie S, Grant D, Indrevoll B, Smeets R, von Ahsen O, Kristian A, Lejeune P, Hennekes H, Karlsson J, Bjerke RM, Ryan OB, Cuthbertson AS, Mumberg D. Preclinical Efficacy of a PSMA-Targeted Thorium-227 Conjugate (PSMA-TTC), a Targeted Alpha Therapy for Prostate Cancer. Clin Cancer Res. 2020 Apr 15;26(8):1985-1996. doi: 10.1158/1078-0432.CCR-19-2268. Epub 2019 Dec 12. PMID 31831560